CLINICAL TRIAL: NCT03802786
Title: An Open-label, Single-dose, Parallel-group Study to Assess the Pharmacokinetics of Imeglimin in Subjects With Moderate Hepatic Impairment Compared to Matched Healthy Control Subjects
Brief Title: Pharmacokinetics of Imeglimin in Hepatic Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXL008-024
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hepatic Impairment
Keywords: pharmacokinetics
MeSH Terms: interventions — imeglimin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate hepatic impairment (Experimental): Single dose of Imeglimin
  Interventions: Drug: Imeglimin
- Normal hepatic function (Experimental): Single dose of Imeglimin
  Interventions: Drug: Imeglimin

INTERVENTIONS:
Drug: Imeglimin — Single administration dose of imeglimin

SUMMARY:
This is a Phase 1, single-centre, open-label, parallel-group study in subjects with moderate hepatic impairment and subjects with normal hepatic function. Child-Pugh (CP) scoring will be used to determine hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* BMI :18.0 and 40.0 kg/m2 and weight ≥50 kg.
* Stable hepatic impairment or normal hepatic function for healthy volunteer
* No clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, and clinical laboratory evaluations (Subjects with moderate hepatic impairment may have medical findings consistent with their hepatic dysfunction)
* Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception
* Informed consent signature

Exclusion Criteria:

* Clinically relevant abnormal findings at the screening assessment
* Severe adverse reaction to any drug or sensitivity to the trial medication or its componentsClinically significant vital signs outside the acceptable range at screening
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Drug or alcohol abuse
* Positive test HIV
* Smoking more than 10 cig/day
* Participation in other clinical trials of unlicensed or prescription medicines

Exclusion criteria for healthy volunteer

* Positive test for HBV, HBC
* eGFR less than 90 mL/min/1.73 m2
* liver diseases

Exclusion criteria for hepatic impaired

* eGFR less than 80 mL/min/1.73 m2
* Hepatic impairment due to non liver disease
* History of hepatocellular carcinoma or acute liver disease
* CLinically significant change in liver disease status within 6 months
* ascites
* encephalopathy grade III or IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
PK parameters of imeglimin | At Day 1
  Cmax: peak plasma concentration after dosing

SECONDARY OUTCOMES:
PK parameters of imeglimin | From day 1 to day 2
  AUC last:area under the concentration-time curve
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From day 1 to day 7
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Chevalier, Study Director — Poxel SA
Locations (1):
- Apex, Munich, Germany